CLINICAL TRIAL: NCT01501513
Title: A Safety, Tolerance and Efficacy Evaluation of 3 Different Bowel Cleansing Preparations in Adult Subjects, Including the Elderly and Subjects With Hepatic or Renal Insufficiency
Brief Title: A Safety Study of 3 Different Bowel Cleansing Preparations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BLI800-440
Record Dates: First submitted 2011-12-22; First posted 2011-12-29 (Estimated); Results first posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Colonoscopy; Bowel Preparation; Endoscopy
Keywords: colonoscopy; bowel preparation; endoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BLI800 approved preparation regimen (Experimental): BLI800 approved preparation regimen
  Interventions: Drug: BLI800 approved preparation regimen
- BLI800 investigational preparation regimen (Experimental): BLI800 investigational preparation regimen
  Interventions: Drug: BLI800 investigational preparation regimen
- PEG-3350 based bowel preparation (Active Comparator): PEG-3350 based bowel preparation
  Interventions: Drug: PEG-3350 based bowel preparation

INTERVENTIONS:
Drug: PEG-3350 based bowel preparation — solution for oral administration prior to colonoscopy
  Arms: PEG-3350 based bowel preparation
Drug: BLI800 approved preparation regimen — solution for oral administration prior to colonoscopy
  Arms: BLI800 approved preparation regimen
Drug: BLI800 investigational preparation regimen — solution for oral administration prior to colonoscopy
  Arms: BLI800 investigational preparation regimen

SUMMARY:
The objective of this study is to compare the safety, tolerance and efficacy of BLI800 (approved and investigational regimens) to an approved control preparation as bowel preparations prior to colonoscopy in adult patients, particularly including the elderly and those with renal and/or hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients who are undergoing colonoscopy for a routinely accepted indication.
* At least 18 years of age
* If female, and of child-bearing potential, is using an acceptable form of birth control
* Negative urine pregnancy test at screening, if applicable
* In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Exclusion Criteria:

* Subjects with known or suspected ileus, severe ulcerative colitis, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis or megacolon.
* Subjects who had previous significant gastrointestinal surgeries.
* Subjects who have uncontrolled clinically significant pre-existing electrolyte disturbances.
* Subjects with severe liver or renal insufficiency.
* Subjects with a history of congestive heart failure or other clinically significant cardiac abnormality.
* Subjects with impaired consciousness that predisposes them to pulmonary aspiration.
* Subjects undergoing colonoscopy for foreign body removal and decompression.
* Subjects who are pregnant or lactating, or intending to become pregnant during the study.
* Subjects of childbearing potential who refuse a pregnancy test.
* Subjects allergic to any preparation components
* Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures.
* Subjects who have participated in an investigational surgical, drug, or device study within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03-04 (Actual); Study Completion 2013-03-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - University of South Alabama, Mobile, Alabama
  - Advanced Clinical Research Institute, Anaheim, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Miami Research Associates, South Miami, Florida
  - Indiana University, Indianapolis, Indiana
  - Delta Research Partners, Monroe, Louisiana
  - Commonwealth Clinical Studies, Brockton, Massachusetts
  - Gastrointestinal Associates, Jackson, Mississippi
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - Carolina Digestive Health Associates, Charlotte, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Northwest Gastroenterology, Portland, Oregon
  - ClinSearch, Chattanooga, Tennessee
  - Franklin Gastroenterology, Franklin, Tennessee
  - Charlottesville Medical Research, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BLI800 Approved Preparation Regimen | BLI800 Investigational Preparation Regimen | PEG-3350 Based Bowel Preparation
Started | 184 | 180 | 177
Completed | 168 | 165 | 164
Not Completed | 16 | 15 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BLI800 Approved Preparation Regimen | BLI800 Investigational Preparation Regimen | PEG-3350 Based Bowel Preparation | Total
Number analyzed (Participants) | 184 | 180 | 177 | 541
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (11.5) | 57.6 (10.2) | 56.6 (10.9) | 57.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 107 | 111 | 319
  Male | 83 | 73 | 66 | 222
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 19 | 18 | 52
  Not Hispanic or Latino | 169 | 161 | 159 | 489
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 4 | 3 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 24 | 20 | 31 | 75
  White | 156 | 156 | 139 | 451
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 184 | 180 | 177 | 541

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Successful Bowel Preparation
Description: Successful bowel preparation is defined as a preparation rated as Excellent or Good by the blinded endoscopist on a 4 point scale (Excellent, Good, Fair, Poor).
Time Frame: Day of colonoscopy
Population: The Primary Efficacy Outcome includes all patients that took a portion of study preparation, except those that did not undergo colonoscopy for a reason other than safety or efficacy (e.g., patient could not get a ride to their colonoscopy).
Measure: Count of Participants; unit: Participants
Arm/Group | BLI800 Approved Preparation Regimen | BLI800 Investigational Preparation Regimen | PEG-3350 Based Bowel Preparation
Number analyzed (Participants) | 183 | 179 | 177
Participants | 175 | 132 | 137
Statistical Analysis 1: Comparison: BLI800 Approved Preparation Regimen vs BLI800 Investigational Preparation Regimen vs PEG-3350 Based Bowel Preparation; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Count and Percentage of Subjects With Adverse Events Through Day of Colonoscopy
Description: Count and Percentage of subjects with AEs through Day of Colonoscopy based on 3% threshold. Outcome measure time frame represents the day prior to colonoscopy (when preparation Dose 1 is taken) and the day of colonoscopy (when preparation Dose 2 is taken).
Time Frame: 2 days
Population: All subjects that took any portion of study preparation.
Measure: Count of Participants; unit: Participants
Arm/Group | BLI800 Approved Preparation Regimen | BLI800 Investigational Preparation Regimen | PEG-3350 Based Bowel Preparation
Number analyzed (Participants) | 184 | 180 | 177
Participants
  Abdominal distension | 79 | 75 | 83
  Abdominal pain | 65 | 56 | 50
  Nausea | 77 | 50 | 54
  Vomiting | 14 | 18 | 13
  Discomfort | 105 | 92 | 90
  Anion gap increased | 9 | 6 | 4
  Headache | 6 | 7 | 11

3. Secondary Outcome: Count and Percentage of Subjects With Adverse Events After Colonoscopy Through Follow-up Day 7
Description: Count and Percentage of subjects with AEs reported after colonoscopy through follow-up Day 7 based on 3% threshold. Outcome measure time frame represents the period following colonoscopy through follow-up Day 7 (7 days).
Time Frame: 7 days
Population: All subjects who took a portion of study preparation.
Measure: Count of Participants; unit: Participants
Arm/Group | BLI800 Approved Preparation Regimen | BLI800 Investigational Preparation Regimen | PEG-3350 Based Bowel Preparation
Number analyzed (Participants) | 184 | 180 | 177
Participants
  Nausea | 3 | 11 | 7
  Abdominal distension | 10 | 18 | 25
  Abdominal pain | 11 | 10 | 11

ADVERSE EVENTS:
Time Frame: 6 months
Description: The Serious Adverse Event and All-Cause Mortality tables reflect all SAEs and deaths which occurred during the study. The Other Adverse Events table reflect all adverse events that occurred during the study.
Arm/Group | BLI800 Approved Preparation Regimen | BLI800 Investigational Preparation Regimen | PEG-3350 Based Bowel Preparation
All-Cause Mortality (participants affected / at risk) | 0/184 | 1/180 | 0/177
Serious Adverse Events (participants affected / at risk) | 4/184 | 12/180 | 3/177
Other Adverse Events (participants affected / at risk) | 145/184 | 129/180 | 127/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLI800 Approved Preparation Regimen (N=184) | BLI800 Investigational Preparation Regimen (N=180) | PEG-3350 Based Bowel Preparation (N=177)
Worsening of vague upper abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Splenic injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bilateral silicone breast implant rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lower anterior resection of the rectum (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Acute renal failure (post-operative) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bilateral breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bilateral mastectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Left breast tissue expander removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Sigmoid colon resection (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Laparoscopic assisted anterior rectosigmoid colon resection (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Septic shock secondary to cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Coffee ground emesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Melena (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cirrhosis - Liver transplant (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Surgery for sigmoid colectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Colon resection (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Attenuated familial adenomatous polyposis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Stage II breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Worsening of re-current diabetic left ankle ulceration (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hospitalization from severe anemia due to vaginal bleed (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Hospitalization for chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BLI800 Approved Preparation Regimen (N=184) | BLI800 Investigational Preparation Regimen (N=180) | PEG-3350 Based Bowel Preparation (N=177)
Abdominal distension (Gastrointestinal disorders) | 84 | 89 | 94
Abdominal pain (Gastrointestinal disorders) | 71 | 65 | 55
Nausea (Gastrointestinal disorders) | 81 | 61 | 56
Vomiting (Gastrointestinal disorders) | 16 | 23 | 16
Discomfort (General disorders) | 108 | 100 | 95
Headache (Nervous system disorders) | 7 | 8 | 12
Urinary tract infection (Infections and infestations) | 10 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sole disclosure restriction which sponsor imposes on the PI is a sixty (60) day limited restriction in order to the protect potentially proprietary information which may be patentable.